CLINICAL TRIAL: NCT05158582
Title: Comparison of Conventional Exercise Protocols and Specific Modified Exercise Program for Low Back Pain in Racketlon Players
Brief Title: Specific Modified Exercise Program for Low Back Pain in Racketlon Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01018 Zainab Saad
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPECIFIC MODIFIED EXERCISE PROGRAM GROUP (Experimental): The modified exercise group will perform 12 exercises.
  Interventions: Other: SPECIFIC MODIFIED EXERCISE PROGRAM GROUP
- CONVENTIONAL EXERCISES PROGRAM GROUP (Active Comparator): The conventional exercises program will perform conventional exercises.
  Interventions: Other: CONVENTIONAL EXERCISES PROGRAM GROUP

INTERVENTIONS:
Other: SPECIFIC MODIFIED EXERCISE PROGRAM GROUP — The modified exercise program group will perform following exercises:
  Resisted static Squats SLER Banded rows SL Banded Jumps Resisted explosive reverse lunges 5hurdle Jumps Elevated single leg Swiss ball Bosu Banded Stars RLE Barbell lunge Static shoulder Abd.with banded leg Add Ant.Banded static squat with medball press Bosu banded superman Sit ups
  Arms: SPECIFIC MODIFIED EXERCISE PROGRAM GROUP
Other: CONVENTIONAL EXERCISES PROGRAM GROUP — The conventional exercise program group will perform the same exercises as they doing for their low back pain.
  Arms: CONVENTIONAL EXERCISES PROGRAM GROUP

SUMMARY:
To compare the effects of conventional exercise protocol and specific modified exercise program to prevent low back pain in racketlon players.

DETAILED DESCRIPTION:
Racketlon is a combination sport in which competitors play a sequence of the four most popular racket sports: Table Tennis, Badminton, squash and tennis. Squash (racquet sport) is an intermittent high-intensity competitive racquet sport that requires quick movements as maintaining control over the placement of the ball with the greatest spatial awareness that is played globally through racquet sports are enjoyed throughout the world and are increasing in their popularity. Since this game encumbers a high level of fitness from the players, who are usually active for the majority of the playing time. Squash players are physically challenged as they are engaged in continuous repetitive training and frequent participation in game to improve their fitness and skills.

The purpose of this study is to find the effects of modified exercise program on LBP in racketlon players. The modified exercise program is a 5-Week Linear Periodization Program, which had effects on Maximal Strength and Speed on elite squash players. This study will find whether this 5-week linear periodization program has an effect to prevent low back pain in racketlon players.

ELIGIBILITY:
Inclusion Criteria:

* Active Male Racketlon player involved in sport activities for at least 3 times per week
* Age between 20-30 years.
* Players having ≥ 2 episodes of mechanical low back pain in past 6 months.

Exclusion Criteria:

Any upper and lower limb injury.

* History of metabolic diseases.
* History of recent fractures.
* History of spinal radiculopathy

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Micheli functional scale (MFS): | 5 weeks
  The Micheli functional scale (MFS) was developed as a back-specific tool for functional assessment in young athletes. This scale is a brief and reliable rating scale to quantify pain intensity and athletic function and determines the degree of the back pain associated with sports activity limitations, back extension/or upright activities, sitting/or flexion activities, and jumping activity. The MFS is a self-report questionnaire and contains 5 items consisting of a symptom question, 3 activity-related questions, and a visual analogue scale (VAS) for pain intensity. The total score is calculated by adding questionnaire responses (range 0 - 15) plus VAS score (range 0 - 10). This maximum total score of 25 is then multiplied by 4. The range of total scores is from 0 (least amount of difficulty) to 100 (the most amount of difficulty).
1 Minute Push-up Test (PUT): | 5 Weeks
  The test began with the athlete in a push-up position, hands placed shoulder width apart with elbows in full extension. The athlete was asked to maintain a neutral spine throughout the movement. A 4-inch block was positioned directly below the athletes' chests to standardize push up depth every time. 1 repetition was counted when the athlete performs a push up and the chest comes into contact with the block and then returning to the starting position. Each athlete was given 1 minute to perform a maximum number of repetitions.
Kraus -Weber Test for lower back muscles | 5 Weeks
  The Kraus-Weber Test involves a series of tests that measure minimum strength & flexibility of the back, abdominals, psoas, and hamstring muscles. The Kraus-Weber fitness test protocols, a series of six medical fitness tests measuring the strength and flexibility of key postural (core) muscles. This abdominal test assesses the strength of the abdominal and psoas muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, Ph.D*, Principal Investigator — Riphah International University
Locations (1):
- Safari Sports Club, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No